CLINICAL TRIAL: NCT05291598
Title: IV Meloxicam for Pain Management Post TJA: Prospective Randomized Trial
Brief Title: Meloxicam for Pain Management After Total Joint Arthroplasty (TJA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Victor Hugo Hernandez, Professor Chief - Division of Arthroplasty & Adult Reconstruction, Department of Orthopaedics, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20211214
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Total Knee Replacement; Total Hip Replacement
MeSH Terms: interventions — Meloxicam; Ketorolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac group (Active Comparator): Participants will receive the institution specific joint replacement pain protocol, including ketorolac.
  Interventions: Drug: Ketorolac
- IV meloxicam group (Experimental): Participants will receive the institution specific joint replacement pain protocol, however with IV meloxicam substituted for ketorolac.
  Interventions: Drug: IV meloxicam

INTERVENTIONS:
Drug: IV meloxicam — Participants will be administered meloxicam 30 mg IV push pre-operatively.
  Arms: IV meloxicam group
Drug: Ketorolac — Participants will be treated with ketorolac 15 mg IV push intra-operatively, followed by 15 mg IV push every 6 hours scheduled for 2 doses.
  Arms: Ketorolac group

SUMMARY:
The purpose of this project is to determine if a change in patient reported pain, nausea and vomiting after total knee and hip arthroplasty could be observed with the substitution of Intravenous meloxicam for ketorolac in the current established peri-operative pain protocol and if these changes lead to a decrease in opioid consumption (in morphine equivalents).

ELIGIBILITY:
Inclusion Criteria:

1. Patients over the age of 18,
2. Patients undergoing primary total knee or primary total hip replacement at the University of Miami Hospital,
3. Patients that have capacity to provide medical consent

Exclusion Criteria:

1. All patients under the age of 18
2. Prisoners, diabetics, increased risk of bleeding, and pregnant women.
3. Patients with prior surgery or history of infection on the joint of interest.
4. Patients with an estimated glomerular filtration rate (eGFR) <50 ml/min
5. Patients on dialysis or renal transplant.
6. Patients on steroid preoperatively.
7. Allergy to sulfas
8. Inability to provide medical consent.
9. Any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements will exclude the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor H Hernandez, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizzo MG, Costello JP 2nd, Constantinescu DS, Samineni AV, Moore MR, Shittu AT, Tabibi O, Osman BM, Fiala RS, D'Apuzzo MR, Hernandez VH. Intravenous Meloxicam Versus Ketorolac for Pain Control Following Total Joint Arthroplasty: A Double-Blind Randomized Controlled Trial. J Arthroplasty. 2025 Oct 28:S0883-5403(25)01331-2. doi: 10.1016/j.arth.2025.10.052. Online ahead of print. PMID 41167538

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketorolac Group: Participants will receive the institution specific joint replacement pain protocol.
  Institution specific joint replacement pain protocol: Participants will be treated with a standard orthopaedic joint replacement protocol which includes:
  * Dexamethasone
  * Tylenol
  * Lyrica
  * Celebrex
  * Meloxicam
  * Oxycodone
  Ketorolac: Participants will be treated with ketorolac 15 mg IV push intra-operatively, followed by 15 mg IV push every 6 hours scheduled for 2 doses.
- IV Meloxicam Group: Participants will be given IV meloxicam for pain management post total knee and hip arthroplasty.
  Institution specific joint replacement pain protocol: Participants will be treated with a standard orthopaedic joint replacement protocol which includes:
  * Dexamethasone
  * Tylenol
  * Lyrica
  * Celebrex
  * Meloxicam
  * Oxycodone
  IV meloxicam: Participants will be administered meloxicam 30 mg IV push pre-operatively.
Period: Overall Study
Arm/Group | Ketorolac Group | IV Meloxicam Group
Started | 114 | 109
Completed | 114 | 109
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketorolac Group | IV Meloxicam Group | Total
Number analyzed (Participants) | 114 | 109 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.65 (9.56) | 64.34 (8.93) | 64.50 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 60 | 122
  Male | 52 | 49 | 101
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.73 (5.49) | 31.10 (5.91) | 30.91 (5.69)
Laterality [Count of Participants; unit: Participants]
  Right | 57 | 58 | 115
  Left | 56 | 51 | 107
  Bilateral | 1 | 0 | 1
Procedure [Count of Participants; unit: Participants]
  Total Hip Arthroplasty | 45 | 44 | 89
  Total Knee Arthroplasty | 69 | 65 | 134
Apfel Score for Postoperative Nausea and Vomiting [Mean (Standard Deviation); unit: units on a scale] — Apfel scores range from 0 to 4, where the higher the score, the greater the predicted 24-h risk of PONV.
  units on a scale | 1.78 (0.90) | 2.00 (0.89) | 1.88 (0.90)

OUTCOME MEASURES:

1. Primary Outcome: Pain Measured by the Numeric Rating Scale
Description: A numeric pain rating scale will be used - a higher pain score would indicate higher pain levels. It is scaled from 0-10.
Time Frame: 2 hours postoperatively
Population: 15 patients in the ketorolac group and 24 in the Meloxicam group did not return survey data in the time period analyzed for this variable and were thus excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 99 | 85
units on a scale | 3.34 (3.25) | 3.32 (3.39)

2. Primary Outcome: Pain Measured by the Numeric Rating Scale
Description: A numeric pain rating scale will be used - a higher pain score would indicate higher pain levels. It is scaled 0-10.
Time Frame: 24 hours postoperatively
Population: 20 patients in the ketorolac group and 25 in the Meloxicam group did not return survey data in the time period analyzed for this variable and were thus excluded.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 94 | 84
units on a scale | 4.06 (3.07) | 3.75 (3.19)

3. Secondary Outcome: Nausea Score as Measured by a Likert Scale
Description: Patients select a score to indicate the severity of their nausea. Scores of 0, 1-2, 3-6, and 7-9 indicate no nausea, mild nausea, moderate nausea, and severe nausea, respectively. The score 10 is assigned to vomiting.
Time Frame: 2 hours postoperatively
Population: 16 patients in the ketorolac group and 24 in the Meloxicam group did not return survey data in the time period analyzed for this variable and were thus excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 98 | 85
score on a scale | 0.42 (1.62) | 0.54 (1.80)

4. Secondary Outcome: Nausea Score as Measured by a Likert Scale
Description: as for outcome 3
Time Frame: 24 hours postoperatively
Population: 21 patients in the ketorolac group and 26 in the Meloxicam group did not return survey data in the time period analyzed for this variable and were thus excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 93 | 83
score on a scale | 0.48 (1.53) | 0.29 (0.96)

5. Secondary Outcome: Length of Stay as Measured by Hours in the Hospital
Description: Length of stay for the patient as measured in hours from surgery until the moment of discharge
Time Frame: Until patient discharged from the hospital
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 114 | 109
hours | 37.87 (49.81) | 41.56 (34.30)

6. Secondary Outcome: Length of Stay as Measured by Hospital Nights
Description: The total number of overnights spent in the hospital between surgery and discharge
Time Frame: From surgery until discharge
Measure: Mean (Standard Deviation); unit: nights
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 114 | 109
nights | 1.51 (2.07) | 1.63 (1.40)

7. Secondary Outcome: Length of Stay as Measured by Same Day Discharges
Description: The number of patients which were able to be discharged home the same day as their surgical procedure
Time Frame: From surgery until discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 114 | 109
Participants | 23 | 10

8. Secondary Outcome: Opioid Consumption as Measured by Morphine Milligram Equivalents (MME)
Description: The amount of opioids a patient consumes converted into MME for standard comparisons
Time Frame: Within 2 hours postoperatively
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 114 | 109
morphine milligram equivalents | 1.98 (4.84) | 2.00 (3.09)

9. Secondary Outcome: Opioid Consumption as Measured by Morphine Milligram Equivalents (MME)
Description: The amount of opioids a patient consumes converted into MME for standard comparisons
Time Frame: Within 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 114 | 109
morphine milligram equivalents | 20.59 (26.46) | 28.21 (24.22)

10. Secondary Outcome: Renal Injury as Measured by the Change in Creatinine Levels
Description: The change in creatinine levels per patient as by comparing their standard preoperative lab creatinine values with the standard postoperative lab creatinine values before discharge from the hospital after their procedure, up to 1 week postoperatively.
Time Frame: From preoperative baseline labs while hospitalized, up to 1 week
Population: 28 patients in the ketorolac group and 24 in the Meloxicam group did not have available data in the time period analyzed for this variable and were thus excluded. Both Arm/Groups had the same reporting identical values.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ketorolac Group | IV Meloxicam Group
Number analyzed (Participants) | 86 | 85
mg/dL | 0.09 (0.19) | 0.09 (0.19)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Ketorolac Group | IV Meloxicam Group
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/109
Other Adverse Events (participants affected / at risk) | 0/114 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT05291598/Prot_SAP_001.pdf